CLINICAL TRIAL: NCT06343311
Title: An Open-Label, Dose Escalation, Multi-Center Phase I/II Clinical Trial of EB103 T-Cell Therapy in Adults With Relapsed/Refractory (R/R) B-Cell Non-Hodgkin's Lymphoma (NHL)
Brief Title: T-Cell Therapy (EB103) in Adults With Relapsed/Refractory B-Cell Non-Hodgkin's Lymphoma (NHL)
Acronym: STARLIGHT-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Estrella Biopharma, Inc. (Industry)
Collaborators: Eureka Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Organization: Estrella Immunopharma, Inc. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EBUS22CD19AR100
Record Dates: First submitted 2024-03-14; First posted 2024-04-02 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: B-Cell Non-Hodgkin's Lymphoma (NHL); Lymphoma, Non-Hodgkins; Lymphomas Non-Hodgkin's B-Cell; Non-Hodgkin Lymphoma; Non-Hodgkin's Lymphoma; Large B-Cell Lymphoma; Lymphoma, Non-Hodgkin's, Adult; Lymphoma; Refractory Non-Hodgkin Lymphoma; Relapsed Non-Hodgkin Lymphoma; Lymphoma, Non-Hodgkin; HIV Associated Lymphoma; CNS Lymphoma; High-grade B-cell Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma
Keywords: B-Cell Non-Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; NHL; Lymphoma; Large B-Cell Lymphoma; Refractory Non-Hodgkin Lymphoma; Relapsed Non-Hodgkin Lymphoma; HIV Lymphoma; CNS Lymphoma; High-grade B-cell Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma; Lymphoma, Primary Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EB103 (Other): Approximately six (6) subjects will be treated to determine the RP2D. At the designated RP2D, approximately fifteen (15) additional subjects will be treated.
  Interventions: Biological: EB103

INTERVENTIONS:
Biological: EB103 — EB103 is an autologous T-cell therapy whereby a subject's own T cells are transduced with a lentiviral vector expressing the EB103 transgene.

SUMMARY:
This is an open-label, dose escalation, multi-center, Phase I/II clinical trial to assess the safety of an autologous T-cell therapy (EB103) and to determine the Recommended Phase II Dose (RP2D) in adult subjects (≥ 18 years of age) who have relapsed/refractory (R/R) B-cell NHL. The study will include a dose escalation phase followed by an expansion phase.

DETAILED DESCRIPTION:
This is an open-label, dose escalation, multi-center, Phase I/II clinical trial to assess the safety of EB103 and determine the RP2D in adult subjects (≥ 18 years of age) who have R/R B-cell NHL.

The study will include a dose escalation phase followed by an expansion phase. A traditional dose escalation model (3+3 design) will be used to determine the RP2D, and once determined, the expansion phase will commence. Additional subjects will be enrolled in the expansion phase to further confirm the safety profile of EB103 at the RP2D and evaluate the preliminary efficacy of EB103.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at the time of informed consent
* Histologically confirmed R/R B-cell non-Hodgkin's lymphoma (NHL)
* Adequate organ function
* Relapsed or refractory (R/R) disease defined as ONE OR MORE of the following:

  * R/R after ≥ 2 lines of systemic therapy

    * For the following NHL types: Burkitt lymphoma, Precursor B-cell lymphoblastic lymphoma, or Mantle cell lymphoma: R/R after ≥ 1 lines of systemic therapy
  * Disease progression or recurrence ≤ 12 months after autologous hematopoietic stem cell transplantation (HSCT)
  * For subjects who are considered transplant-ineligible: progressive disease as best response after ≥ 4 cycles of first-line therapy and stable disease as best response after ≥ 2 cycles of second-line (salvage) therapy; subject must have received an anti-CD20 monoclonal antibody and an anthracycline as one of their qualifying regimens
* All subjects must have received an appropriate chemoimmunotherapy regimen which at a minimum includes an:

  * Anti-CD20 monoclonal antibody AND
  * An anthracycline-containing chemotherapy regimen
* Positron emission tomography (PET)-positive disease according to Cheson 2014
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Toxicities due to prior therapy must be stable and recovered to Grade 1 or less

Exclusion Criteria:

* Prior CD19-targeted cellular therapy
* History of Richter's transformation of chronic lymphocytic leukemia (CLL)
* History of another primary malignancy that has not been in remission for ≥ 2 years.
* History or presence of clinically relevant Central Nervous System (CNS) pathology
* CNS disease which is progressing on most recent therapy or with a parenchymal mass which is likely to cause clinical symptoms
* Subjects with active cardiac lymphoma involvement which is not responding to treatment
* History of myocardial infarction, cardiac angioplasty and stenting, unstable angina, or other clinically significant cardiac disease within 6 months of informed consent
* Active, uncontrolled systemic bacterial, fungal, or viral infection. Patients with HIV, hepatitis B, or hepatitis C are eligible provided their infection is being treated and the viral load is controlled.
* History of autoimmune disease resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years
* History of severe, immediate hypersensitivity reaction to any agents used in this study, including the conditioning chemotherapeutic agents
* Venous thrombosis or embolism not managed on a stable regimen of anticoagulation
* Autologous HSCT within 3 months of informed consent
* Subjects with a prior allogeneic transplant at least 6 months prior to study enrollment are eligible unless experienced graft-versus-host disease (GvHD) that requires ongoing treatment with systemic steroids or other systemic GvHD therapy, such as a calcineurin inhibitor, within 12 weeks of initial screening
* Live vaccine within 3 months prior to planned start of conditioning regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the Dose Limiting Toxicities of EB103. | Time Frame: 28 days
  The incidence of Dose Limiting Toxicities (DLTs) that occur within 28 days following EB103 T-cell infusion will be assessed. A DLT consists of any adverse event (AE) or abnormal laboratory value assessed as unrelated to disease, disease progression, concomitant medication, or intercurrent illness that occurs within 28 days following EB103 T-cell infusion and meets specified criteria as outline in the clinical protocol. The type, frequency, and severity of each DLT, AE, and abnormal laboratory value will be documented to assess the safety and tolerability of EB103.
Incidence rates of Treatment-Emergent Adverse Events of EB103. | Time Frame: 90 days
  The type, frequency, and severity of Treatment-Emergent Adverse Events (TEAEs) will be assessed and includes an AE that starts any time from initiation of EB103 administration through and including 90 days after EB103 administration.
  Listing and summaries will be prepared for the following type of events: TEAEs, SAEs, Grade 3 or higher AEs, treatment related AEs (conditioning chemotherapy, protocol-mandated procedures, or EB103), and AEs leading to death. AESIs, including but not limited to acute infusion reaction, CRS, ICANS, prolonged cytopenia, TLS, MAS/HLH, SPM, and hypogammaglobulinemia.
Incidence rates Treatment-Emergent Laboratory Abnormalities reported for EB103. | Time Frame: 90 days
  The type, frequency, and severity after Treatment-Emergent Laboratory Abnormalities will be assessed and includes a laboratory abnormality that, compared to baseline, worsens by at least one grade with 90 days after EB103 administration.
To determine the Recommended Phase II Dose (RP2D) of EB103. | Time Frame: 21 months
  The RP2D will be determined by the study Dose Escalation Committee (DEC) and chosen based on the maximum tolerated dose (MTD) but will not exceed the MTD and the maximum administered dose (MAD). The RP2D will also be based on the manufacturing capability.

SECONDARY OUTCOMES:
To assess the Overall Response Rate of EB103 in our study subject population. | Time Frame: Up to 2 years
  The Overall Response Rate (ORR), defined as the proportion of subjects with a Best Overall Response (BOR) of either Complete Response (CR) or Partial Response (PR) will be assessed.
To assess the Disease Control Rate of EB103 in our study subject population. | Time Frame: Up to 2 years
  The Disease Control Rate (DCR), defined as the proportion of subjects with BOR of either Complete Response (CR), Partial Response (PR), or Stable Disease (SD) will be assessed.
To assess the Duration of Response of EB103 in our study subject population. | Time Frame: Up to 2 years
  The Duration of Response (DOR), defined as the time from first response to Progressive Disease (PD) or death will be assessed.
To assess the Progression-Free Survival rate of EB103 in our study subject population. | Time Frame: Up to 2 years
  The Progression-Free Survival (PFS), defined as the time from EB103 infusion to PD or death will be assessed.
To assess the Event-Free Survival rate of EB103 in our study subject population. | Time Frame: Up to 2 years
  The Event-Free Survival (EFS) will be defined as the time from EB103 T-cell infusion to the earliest of the following events: death from any cause, PD, or starting a new anticancer therapy.
To assess the Overall Survival rate of EB103 in our study subject population. | Time Frame: Up to 2 years
  The Overall Survival (OS) will be defined as the time from EB103 T-cell infusion to the date of death.
To characterize the pharmacokinetic (PK) profile of EB103 by measuring the peak exposure (Cmax). | Time Frame: Up to 2 years
  The peak exposure (Cmax) will be measured in our study subject population.
To characterize the pharmacokinetic (PK) profile of EB103 by measuring the time to reach peak exposure (Tmax). | Time Frame: Up to 2 years
  Time to reach peak exposure (Tmax) will be measured in our study subject population.
To characterize the pharmacokinetic (PK) profile of EB103 by measuring the partial area under the curve (pAUC). | Time Frame: Up to 2 years
  Partial area under the curve (pAUC) will be measured in our study subject population.

CONTACTS AND LOCATIONS:
Overall Officials: Pei Wang, PhD, Study Director — Eureka Therapeutics Inc.
Locations (2):
- United States (2):
  - University of California, Davis, Sacramento, California
  - Baylor Scott & White Research Institute, Texas Oncology, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No